CLINICAL TRIAL: NCT04610606
Title: A Novel Multimodal Intervention for Surgical Prehabilitation of Patients With Lung Cancer: Pilot Study
Brief Title: Pilot Prehabilitation Intervention in Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: McGill University (Other)
Collaborators: Peri-Operative Program Charitable Foundation (Unknown); MUHC-Montreal General Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Stéphanie Chevalier, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUHC REB 2020-5633
Record Dates: First submitted 2020-09-24; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer; Surgery
Keywords: Prehabilitation; Nutritional supplement
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, controlled trial of two parallel arms: multimodal intervention (MM) and standard of care (SOC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal intervention (MM) (Experimental): Multimodal prehabilitation including structured exercise (1 supervised exercise session per week + home-based exercise program), nutritional optimization (diet + mixed nutrient supplement containing whey protein, leucine, vitamin D and omega 3 fatty acids) and relaxation strategies.
  Interventions: Behavioral: Multimodal intervention (MM)
- Standard of care (SOC) (No Intervention): Education on benefits of physical activity and healthy diet, with no specific information.

INTERVENTIONS:
Behavioral: Multimodal intervention (MM) — Exercise: Moderate intensity resistance and aerobic exercise, including one weekly supervised session and a home-based program. Participants were asked to 1) accumulate 30 min of aerobic exercise per day of their preferred type (ex. walking) and 2) perform 30 min of resistance exercise targeting major muscle groups, every second day for 2 sets of 8-12 reps.
  Nutrition: Optimize diet with protein-rich foods to meet protein intake of >1.2 g/kg/d and energy of 25-30 kcal/kg/d. The supplement consists of whey protein isolate (with the goal of reaching 1.5 g/kg/d, providing 25 g/meal), 6g of leucine, fruit-flavored fish oil added with vitamin D.
  Relaxation strategies: private consultations with psychology-trained personnel whereby techniques aimed at reducing anxiety are practiced. Participants are also provided with a compact disc with relaxation exercises to be used at home 2-3 times per week.
  Arms: Multimodal intervention (MM)

SUMMARY:
Lung cancer is the second most prevalent cancer in Canada and the leading cause of cancer-related mortality worldwide. Patients diagnosed at earlier (non-metastatic) stages are potential candidates for surgical tumor removal. However, they often present with poor nutritional status and physical function adding to the major catabolic stress imposed by surgery that negatively impacts recovery and survival after surgery. The purpose of this study is to investigate the potential benefits of a prehabilitation program that includes a combined nutritional supplement (whey protein, leucine, vitamin D and omega-3 fatty acids) with exercise and relaxation techniques for 4 weeks before surgery and continued for 8 weeks after surgery on functional pre- and postoperative outcomes, versus standard hospital care (control). Investigators will study whether the prehabilitation program improves physical performance, muscle mass and quality of life in patients undergoing lung cancer resection. The specific objective of this pilot study is to test feasibility and adherence to intervention, and generate pilot data to inform the design of a larger trial.

DETAILED DESCRIPTION:
RATIONALE: The preoperative period is an opportune time to actively engage and empower patients in improving their functional, nutritional and mental status in anticipation of the surgical stress. Considering that lung cancer patients often present with poor nutritional status and physical function prior to surgery providing a nutritional supplement to increase protein, leucine, vitamin D and omega-3 FA intake with a structured exercise program and relaxation techniques should improve muscle mass, strength and physical performance.

MAIN OBJECTIVE: to test the effect of a multimodal prehabilitation intervention (MM) combining a mixed-nutrient supplement with structured exercise training against standard of care (SOC), on functional pre- and postoperative outcomes in surgical patients with lung cancer, in an open-label RCT.

The present is a pilot study aiming to generate feasibility data (recruitment rate, compliance, attrition) and preliminary outcome data to support a larger trial.

STUDY DESIGN: Open-label, randomized, controlled trial of two parallel arms: multimodal intervention (MM) and standard of care (SOC). After baseline assessment, patients will be randomized to either group in a 1:2 SOC:MM ratio using a computer-generated randomization scheme by block of four, with stratification by sex and functional capacity (< or > 400 m on the 6MWT). Consecutive adult patients scheduled for elective video-assisted thoracic surgery or open thoracotomy surgery of NSCLC stages I, II or IIIa, will be approached following their first appointment with their surgeon at the MUHC-Montreal General Hospital.

INTERVENTION: The EXP arm will ingest a multi-nutrient supplement consisting of whey protein + leucine and fish oil + vitamin D, perform structured exercise and relaxation techniques for 4 weeks prior to surgery and 8 weeks after surgery. Control group will received standard hospital care and education on benefits of physical activity and healthy diet. Outcome assessment will be performed at baseline, preoperative, 4 and 8 weeks postoperatively.

OUTCOMES: Primary: feasibility; Secondary: physical function, muscle strength, volume and density, body composition, quality of life, length of stay and post-operative complications; Other: dietary intake, physical activity, clinical markers.

STATISTICAL ANALYSIS: This is a pilot study designed to generate data on feasibility and compliance to the intervention and study tests; it is not powered for identifying statistical differences in the main outcomes. The investigators will recruit 36 participants on a 1:2 ratio (12 SOC: 24 MM).

ELIGIBILITY:
Inclusion Criteria:

* adult men and women with NSCLC stages I, II or IIIa, planned for video-assisted thoracic surgery (VATS) or open thoracotomy surgery for cancer resection or exploration.

Exclusion Criteria:

* prior recent (<3 mo) chemotherapy, comorbidities contraindicating exercise (defined as CPET <10 mL O2/kg/min), walking aids other than a cane, glomerular filtration rate <30 mL/min/m2, allergy to milk or seafoods, chronic use of anti-coagulants, hypercalcemia, hypervitaminosis D, insufficient understanding of English or French language to provide informed consent. All medications and co-morbidities will be recorded. Patients taking vitamin D will continue their supplements; risk of potential overdosing will be monitored by serum 25(OH)D levels >80 nmol/L. Those taking n-3 FA supplements will be asked to withhold during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment rate | Over entire recruitment period (approximately 1 year)
  Recruitment rate (measured in percent, compared to expected rates)
Feasibility: Adherence to intervention | Over 12 weeks (4 weeks pre- and 8 weeks post-surgery)
  Adherence to exercise and nutritional interventions (measured in percent, compared to expected rates)
Feasibility: completion of study outcome assessment | Over 12 weeks (4 weeks pre- and 8 weeks post-surgery)
  Completion of study outcome assessments (measured in percent, compared to expected rates)

SECONDARY OUTCOMES:
Functional walking capacity | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Six-minute walking test: measured as the distance walked during 6 minutes, along a 20-m corridor, expressed in m)
Length of hospital stay | 8-week postoperative
  Recorded from medical charts
Post-operative complications | 8-week postoperative
  Recorded from medical charts and will be graded by severity following the Clavien-Dindo classification.
Health related quality of life | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Measured by the cumulative score of the 36-item Short Form Health Survey, score 0-100, higher score means better quality of life.
Quality of Life | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Measured by cumulative score of the Functional Assessment of Cancer Therapy - Lung questionnaires, score 0-136, higher means better quality of life.
Muscle strength - handgrip | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Handgrip strength using hand-held Jamar dynamometer, measured in kg.
Muscle strength - leg | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Isokinetic leg strength (knee extension peak torque) using Biodex, measured in N, on the dominant side.
Muscle volume | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Skeletal muscle volume will be measured in the dominant foreleg, using peripheral quantitative CT (pQCT, Stratec XCT2000).
Muscle radiodensity | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Skeletal muscle density will be measured in the dominant foreleg, using peripheral quantitative CT (pQCT, Stratec XCT2000).
Body composition | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Lean and fat mass will be measured by bioelectrical impedance (InBody 230V)

OTHER OUTCOMES:
Dietary assessment | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Collected using 2 and 3-day food diaries.
Plasma phospholipid n-3 FA profile | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Plasma lipids will be extracted with organic solvents, phospholipids isolated on thin-layer chromatography, and FAs methylated for determination by gas chromatography-flame-ionization analysis. Used as an objective measure of adherence to fish oil.
Serum 25(OH)D | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Concentrations will be measured by the MUHC-Central Lab. Used as an objective measure of adherence to the supplement.
Inflammation | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Will be assessed with serum C-reactive protein (hs-CRP) by MUHC-Central Lab.
Serum albumin | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Will be analyzed as standard procedures by the MUHC-Central Lab.
Pre-albumin | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Will be analyzed as standard procedures by the MUHC-Central Lab.
Hemoglobin | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Will be analyzed as standard procedures by the MUHC-Central Lab.
Exercise tolerance - oxygen consumption | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Assessed using cardiopulmonary exercise testing and measuring oxygen consumption at anaerobic threshold and peak exercise
Exercise tolerance - workload | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Assessed by cardiopulmonary exercise testing at anaerobic threshold and peak exercise
Exercise tolerance - heart rate | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Assessed by cardiopulmonary exercise testing and measured at anaerobic threshold and peak exercise
Pulmonary function (FEV1) | Baseline and 4-week postoperative
  Spirometry standard methods to measure FEV1.
Pulmonary function (FVC) | Baseline and 4-week postoperative
  Spirometry standard methods to measure FVC.
Pulmonary function (FEV1/FVC) | Baseline and 4-week postoperative
  Spirometry standard methods to measure the FEV1/FVC ratio.
Pulmonary function (FEF 25-75%) | Baseline and 4-week postoperative
  Spirometry standard methods to measure FEF 25-75 percent.
Physical activity | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire, score 0 - x (no maximum score), higher mean more activity
Anxiety/depression | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Hospital Anxiety and Depression Scale (questionnaire). Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Nutritional status | Baseline, preoperative, 4-week postoperative and 8-week postoperative
  Patient-Generated Subjective Global Assessment (PG-SGA). In general, the higher total additive scores upon initial exam correlates with more severely malnourished cases (A = well nourished, B = moderately malnourished or suspected malnutrition and C = severely malnourished).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Chevalier, PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
IPD sharing was not planned originally and therefore consent was not obtained for it.

REFERENCES:
- [Derived] Lawson C, Ferreira V, Carli F, Chevalier S. Effects of multimodal prehabilitation on muscle size, myosteatosis, and dietary intake of surgical patients with lung cancer - a randomized feasibility study. Appl Physiol Nutr Metab. 2021 Nov;46(11):1407-1416. doi: 10.1139/apnm-2021-0249. Epub 2021 Jul 15. PMID 34265218